CLINICAL TRIAL: NCT01619761
Title: Natural Killer Cells in Allogeneic Cord Blood Transplantation
Brief Title: NK Cells in Cord Blood Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0493; NCI-2012-02071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0493 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Acute Biphenotypic Leukemia; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukemia in Remission; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; ISS Stage II Plasma Cell Myeloma; ISS Stage III Plasma Cell Myeloma; Myelodysplastic Syndrome; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Lymphocytic Leukemia; Recurrent Hodgkin Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Acute Lymphoblastic Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Small Lymphocytic Lymphoma; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Chronic-Phase; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; fludarabine phosphate; Lenalidomide; Melphalan; Mycophenolic Acid; Rituximab; CT-P10; Tacrolimus; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Plan 1 (NK cells, umbilical cord blood transplant) (Experimental): Patients receive high-dose lenalidomide PO QD on days -8 to -2, fludarabine phosphate IV over 1 hour on days -7 to -4, and melphalan IV over 30 minutes on day -4. CD20 positive patients also receive rituximab IV over 6 hours on days -8 to -4.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Melphalan; Drug: Mycophenolate Mofetil; Biological: Natural Killer Cell Therapy; Biological: Rituximab; Drug: Tacrolimus; Procedure: Umbilical Cord Blood Transplantation
- Treatment Plan 2 (NK cells, umbilical cord blood transplant) (Experimental): Patients receive high-dose lenalidomide PO QD on days -7 to -2, cyclophosphamide IV over 3 hours on day -7, and undergo TBI on day -3. Patients also receive rituximab and fludarabine phosphate as in Treatment Plan 1.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Drug: Mycophenolate Mofetil; Biological: Natural Killer Cell Therapy; Biological: Rituximab; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Procedure: Umbilical Cord Blood Transplantation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic umbilical cord blood transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Treatment Plan 2 (NK cells, umbilical cord blood transplant)
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Treatment Plan 1 (NK cells, umbilical cord blood transplant)
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Biological: Natural Killer Cell Therapy — Given IV
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: Total Body Irradiation; Whole-Body Irradiation
  Arms: Treatment Plan 2 (NK cells, umbilical cord blood transplant)
Procedure: Umbilical Cord Blood Transplantation — Undergo allogeneic umbilical cord blood transplant
  Other Names: Cord Blood Transplantation; UCB transplantation

SUMMARY:
This phase I trial studies the side effects and best way to give natural killer cells and donor umbilical cord blood transplant in treating patients with hematological malignancies. Giving chemotherapy with or without total body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells and natural killer cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility and safety of ex-vivo expanded cord blood (CB) natural killer (NK) cells with double CB transplantation in patients with hematological malignancies.

SECONDARY OBJECTIVES:

I. To monitor engraftment, chimerism, graft versus host disease, and immune reconstitution in patients receiving expanded CB NK cell therapy.

II. To estimate the time to platelet recovery and the time to absolute neutrophil count (ANC) recovery.

III. To estimate overall survival and disease free survival at one year. IV. To study the in-vivo persistence of cord blood NK cells.

OUTLINE:

PREPARATIVE REGIMEN: Patients are assigned to 1 of 2 treatment plans:

TREATMENT PLAN 1: Patients receive high-dose lenalidomide orally (PO) once daily (QD) on days -8 to -2, fludarabine phosphate IV over 1 hour on days -7 to -4, and melphalan IV over 30 minutes on day -4. CD20 positive patients also receive rituximab intravenously (IV) over 6 hours on days -8 to -4.

TREATMENT PLAN 2: Patients receive high-dose lenalidomide PO QD on days -7 to -2, cyclophosphamide IV over 3 hours on day -7, and undergo total body irradiation (TBI) on day -3. Patients also receive rituximab and fludarabine phosphate as in Treatment Plan 1.

NK CELL INFUSION: All patients receive ex-vivo expanded cord blood NK cells IV over 30 minutes on day -2.

TRANSPLANT: All patients undergo allogeneic umbilical cord blood transplant on day 0.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: All patients receive tacrolimus IV or PO on days -2 to 180 followed by taper and mycophenolate mofetil IV over 2 hours or PO thrice daily (TID) on days -3 to 100.

After completion of study treatment, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following hematologic malignancies: acute myelogenous leukemia (AML), induction failure, high-risk for relapse first remission (with intermediate-risk or high-risk cytogenetics, fms-related tyrosine kinase 3 [FLT3] mutation positive and/or evidence of minimal residual disease by flow cytometry), secondary leukemia from prior chemotherapy and/or arising from myelodysplastic syndrome, any disease beyond first remission
* Myelodysplastic syndrome (MDS): primary or therapy related
* Acute lymphoblastic leukemia (ALL): induction failure, primary refractory to treatment (do not achieve complete remission after first course of therapy) or are beyond first remission including second or greater remission or active disease; patients in first remission are eligible if they are considered high risk, defined as any of the following detected at any time: with t(9;22) or t(4;11), hypodiploidy, complex karyotype, secondary leukemia developing after cytotoxic drug exposure, and/or evidence of minimal residual disease, or acute biphenotypic leukemia, or double hit non-Hodgkin's lymphoma
* Non-Hodgkin's lymphoma (NHL) in second or third complete remission, refractory NHL, or relapsed NHL (including relapse post autologous hematopoietic stem cell transplant); double hit lymphomas in first remission or more advanced disease
* Small lymphocytic lymphoma (SLL), or chronic lymphocytic leukemia (CLL) with progressive disease following standard therapy; patients with progressive CLL following standard therapy who meet European Bone Marrow Transplant (EBMT) consensus guidelines of indications for allogeneic stem cell transplantation; this includes patients with (1) lack of response or early relapse within 1 year of receiving a purine analog-containing treatment regimen, (2) disease relapse within 2 years of receiving a purine analog combination therapy or after other therapies such as autologous stem cell transplantation, and (3) CLL associated with tumor protein (p)53 mutations or deletions and/or deletion (del) (17p) requiring therapy; patients must have chemosensitive disease with at least a partial response (PR) or stable disease (SD) with last treatment regimen
* Chronic myeloid leukemia (CML) second chronic phase or accelerated phase
* Hodgkin's disease (HD): induction failures, second or third complete remission, or relapse (including relapse post autologous hematopoietic stem cell transplant)
* Multiple myeloma: stage II or III, symptomatic, secretory multiple myeloma requiring treatment
* Performance score of at least 80% by Karnofsky or 0 to 2 Eastern Cooperative Oncology Group (ECOG)
* Left ventricular ejection fraction greater than 45%
* Pulmonary function test (PFT) demonstrating a diffusion capacity of least 45% predicted
* Creatinine < 1.6 mg/dL
* Serum glutamate pyruvate transaminase (SGPT) =< to 2.0 x normal
* Bilirubin =< to 2.0 x normal
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the Revlimid REMS program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Negative beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 24 months or no previous surgical sterilization and willing to ongoing pregnancy testing while on treatment with lenalidomide
* Woman with child bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide
* Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy
* Patients must have two CB units available which are matched with the patient at 4, 5, or 6/6 human leukocyte antigen (HLA) class I (serological) and II (molecular) antigens; each cord must contain at least 1.5 x 10^7 total nucleated cells/Kg recipient body weight (pre-thaw); cord blood units will be procured through the National Marrow Donor Program (NMDP)
* Have identified a backup cells source in case of engraftment failure; the source can be autologous, related or unrelated
* Patients who have had a prior autologous transplant are eligible

Exclusion Criteria:

* Patients with known history of human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS)
* Active central nervous system (CNS) disease in patient with history of CNS malignancy
* Patients with chronic active hepatitis or cirrhosis; if positive hepatitis serology, the study chair may deem the patient eligible based on the results of liver biopsy
* Patients with known hypersensitivity to lenalidomide and/or rituximab
* Patients who have a matched related donor who is eligible and willing to donate stem cells

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Generation of a minimum of 5 x 10^6 natural killer/kg cells in at least 60% of patients (success rate) | Up to 1 year
  Will be estimated with 90% credible interval.
Treatment-related mortality | 100 days
  The method described by Thall, et al will be used. Will be estimated with 90% credible interval. The product-limit estimator of Kaplan and Meier will be used with 95% confidence intervals.
Incidence of adverse events graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 year
  Changes from baseline in vital signs and laboratory values will be summarized. Tabulate adverse events by severity and relationship to therapy.

SECONDARY OUTCOMES:
Proportion of patients with acute graft-versus-host-disease | Up to 1 year
Proportion of patients with chronic graft-versus-host-disease | Up to 1 year
Overall survival | 1 year
  The product-limit estimator of Kaplan and Meier will be used with 95% confidence intervals.
Disease-free survival | 1 year
  The product-limit estimator of Kaplan and Meier will be used with 95% confidence intervals.
Time to initial platelet recovery | From the infusion of peripheral blood stem cells to the first of 3 consecutive platelet count measurements tested on different days with a count greater than or equal to 20 x 10e9/L, assessed up to 1 year
  Cumulative incidence of platelet recovery will be estimated with the methods of Gooley, et al.
Time to initial absolute neutrophil count recovery | From the infusion of peripheral blood stem cells to the first of 3 consecutive days of an absolute neutrophil count greater than or equal to 0.5 x 10e9/L, assessed up to 1 year
  Cumulative incidence of platelet recovery will be estimated with the methods of Gooley, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Chitra Hosing, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org